CLINICAL TRIAL: NCT06839911
Title: Prevention of Carbapenemase-producing Enterobacteriaceae Epidemics: Evaluation of a Simplified Contact Screening Policy
Brief Title: Prevention of Carbapenemase-producing Enterobacteriaceae Epidemics: Evaluation of a Simplified Contact Screening Policy (CADECO)
Acronym: CADECO
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC25.0003 - CADECO
Record Dates: First submitted 2025-02-11; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Carbapenemase-Producing Enterobacteriaceae

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France, carbapenemase-producing Enterobacteriaceae (CPE) are a significant concern due to their emergence. Efforts to limit their spread focus on reducing antibiotic selection pressure and preventing patient-to-patient transmission. The recommendations issued by the High Council for Public Health in 2010, updated in 2013 and 2019, emphasize the importance of identifying high-risk patients (those who have been hospitalized abroad in the past year) and implementing contact precautions, including single-room isolation and the use of protective clothing. Additional measures include assigning dedicated staff to CPE carriers when possible and conducting systematic weekly screening of all individuals exposed to the same medical or paramedical team, known as contact patient monitoring.

Despite their importance, these recommendations are challenging to implement. Firstly, they require significant resources due to the human and material constraints faced by healthcare systems. Secondly, a large number of contact patients are lost to follow-up and are not screened. The increasing prevalence of CPE carriers has further exacerbated these difficulties.

Epidemic outbreaks, defined by at least one secondary case of CPE carriage among contact patients, require additional control measures. French recommendations for managing an epidemic situation include halting patient transfers between departments, stopping new admissions, and organizing different sectors (CPE carriers, contact patients, and new patients) with dedicated staff for each sector until the outbreak is controlled (with three weeks without a new positive test among contact patients). These measures are even more costly and require time for discussions with hospital management, service reorganization, and hiring additional staff. The difficulties in implementing these measures can have negative effects, such as reduced quality of care and increased staff fatigue.

To address these challenges, some hospitals have adapted their strategies by replacing dedicated teams with a "forward movement" approach and conducting selective screening for only a subset of patients exposed to carriers, based on assessments by infection prevention and control (IPC) specialists. The simplified CPE management protocol was developed in late 2017 at our center. Before that date, French national recommendations for managing carriers and identifying outbreaks were followed. All contacts of a CPE carrier were screened weekly. In 2017, a CPE cohorting unit was implemented at the hospital level for a short period of approximately six months before being discontinued due to difficulties in maintaining continuity of care. In 2018, the selection of a subset of contact patients for screening during each CPE carrier's stay was gradually introduced, without a corresponding change in the definition of an epidemic.

The screening sample is determined by the IPC team based on the duration of contact with the CPE carrier, risk assessment, and geographical proximity. In case of an outbreak, screening is then expanded, and additional measures are implemented as previously described.

This is a retrospective cohort study including adult patients carrying carbapenemase-producing Enterobacteriaceae and comparing stays that resulted in outbreaks to those without outbreaks at Brest University Hospital in the medicine, surgery, or obstetrics departments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient carrying CPE according to HCSP definitions (2010)
* Hospitalized for more than 24 hours at Brest University Hospital in a medicine, surgery, or obstetrics department between 2012 and 2023
* Patient affiliated with a social security system

Exclusion Criteria:

* Patients under legal protection (guardianship, curatorship)
* Deceased patients
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient carrying CPE according to HCSP definitions (2010), hospitalized for more than 24 hours at Brest University Hospital in a medicine, surgery, or obstetrics department between 2012 and 2023
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Detection of a CPE outbreak | untill 2022
  is defined as the identification of CPE with the same resistance enzyme in at least one contact patient of a known carrier.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement